CLINICAL TRIAL: NCT06606665
Title: Comparıson of Balance, Cognıtıve Skılls, Hand Functıons and Qualıty of Lıfe Between Elderly Patıents Wıth Bronchiectasis and Healthy Peers
Brief Title: Balance, Cognıtıve Skılls, Hand Functıons and Qualıty of Lıfe Among Patients with Bronchiectasis and Healthy Peers
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Hilal Denizoğlu Külli, Assoc. Prof., Atlas University
Other Study IDs: IAU-SBE-VHB-01
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Bronchiectasis
Keywords: bronchiectasis; elderly; balance; cognitive ability; hand grip strength; hand functions; quality of life; lower extremity muscle strength; respiratory function parameters; reaction time
MeSH Terms: conditions — Bronchiectasis | interventions — Muscle Strength Dynamometer

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- elderly with bronchiectasis ( EXPERİMENTAL GROUP ): elderly with bronchiectasis
  Interventions:
  Other: Participants will have to sign an informed consent form before the evaluation.
  Demographic information; It will be evaluated with a demographic information evaluation form.
  Other: Cognitive skills; It will be evaluated with the Montreal Cognitive Assessment Scale.
  Other: Reaction time; It will be evaluated with the 12-Red Square Test on the App-coo test application via tablet.
  Other: Quality of life assessment; It will be evaluated with the Nottingham Health Profile.
  Other: Lower extremity muscle strength assessment; It will be evaluated with a 30-second sit-and-stand test.
  Other: Hand grip strength measurement test; It will be evaluated with a dynamometer.
  Other: Pulmonary function assessment; It will be evaluated by spirometry. Other: Balance assessment will be done with the Wii Fit Balance Board.
  Interventions: Other: Cognitive skills test; Other: Reaction time test; Other: Quality of life assessment; Other: Lower extremity muscle strength assessment; Other: Hand grip strength measurement test; Other: Pulmonary function assessment; Other: Balance assessment
- healthy controls (CONTROL GROUP): Age-matched healthy volunteers
  Interventions:
  Other: Participants will have to sign an informed consent form before the evaluation.
  Demographic information; It will be evaluated with a demographic information evaluation form.
  Other: Cognitive skills; It will be evaluated with the Montreal Cognitive Assessment Scale.
  Other: Reaction time; It will be evaluated with the 12-Red Square Test on the App-coo test application via tablet.
  Other: Quality of life assessment; It will be evaluated with the Nottingham Health Profile.
  Other: Lower extremity muscle strength assessment; It will be evaluated with a 30-second sit-and-stand test.
  Other: Hand grip strength measurement test; It will be evaluated with a dynamometer.
  Other: Pulmonary function assessment; It will be evaluated by spirometry. Other: Balance assessment will be done with the Wii Fit Balance Board.
  Interventions: Other: Cognitive skills test; Other: Reaction time test; Other: Quality of life assessment; Other: Lower extremity muscle strength assessment; Other: Hand grip strength measurement test; Other: Pulmonary function assessment; Other: Balance assessment

INTERVENTIONS:
Other: Cognitive skills test — Cognitive skills; It will be evaluated with the Montreal Cognitive Assessment Scale.
  Other Names: MOCA
Other: Reaction time test — Reaction time; It will be evaluated with the 12-Red Square Test on the App-coo test application via tablet.
  Other Names: 12-Red Square Test
Other: Quality of life assessment — Quality of life assessment; It will be evaluated with the Nottingham Health Profile.
  Other Names: NIH
Other: Lower extremity muscle strength assessment — Lower extremity muscle strength assessment; It will be evaluated with a 30-second sit-and-stand test.
  Other Names: 30-second sit-and-stand test
Other: Hand grip strength measurement test — Hand grip strength measurement test; It will be evaluated with a dynamometer.
  Other Names: dynamometer
Other: Pulmonary function assessment — Pulmonary function assessment; It will be evaluated by spirometry.
  Other Names: spirometry
Other: Balance assessment — Balance assessment will be done with the Wii Fit Balance Board.
  Other Names: Wii Fit Balance Board

SUMMARY:
The aim of this study is to comparatively evaluate the parameters of balance, cognitive skills, hand grip strength, reaction time, quality of life and respiratory functions in elderly and healthy peers individuals.

DETAILED DESCRIPTION:
Deterioration of airway patency, respiratory functions, experiencing shortness of breath that limits functional capacity, impairments in health-related quality of life, balance, cognitive skills, hand grip strength and reaction time parameters make physiotherapy approaches important in the treatment of bronchiectasis.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with bronchiectasis and in stable condition,
* No known systemic, orthopedic or neurological disease,
* Can walk,
* Volunteer for research,
* Able to cooperate,
* Elderly individuals aged 65 and over with bronchiectasis
* Healthy elderly individuals aged 65 and over

Exclusion Criteria:

* Individuals under 65 years of age
* Individuals with FEV1 values < 40%
* History of uncontrolled hypertension, arrhythmia and MI in the last month
* Having a history of lung or liver transplantation,
* Unstable angina,
* Those with serious cardiac problems such as advanced heart failure,
* Hemodynamically unstable cases,
* Those who have used antibiotics in the last three weeks,
* Those with acute exacerbation
* Those with insufficient awareness and cooperation,
* Those with pregnancy and malignancy,
* Those who have orthopedic or surgical problems that may prevent tests,
* Those who did not agree to participate in the research

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Elderly with diagnosed with bronchiectasis and age matched healthy volunteers who do not have any diagnosed chronic diseases.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-06-10 (Actual)

PRIMARY OUTCOMES:
Wii Fit Balance Board | The assessment will be administered only once to each participant. All tests will be performed on the same day and will take approximately 30 minutes.
  The use of force platform technologies to assess standing balance is common in a variety of clinical areas. Force platforms can provide detailed quantitative information about underlying movement deficits or postural control mechanisms and responses to sensory manipulations. Force platforms are now considered the gold standard in clinical practice. A reliable and valid study in which the Wii Fit Balance Board can be used as a tool to assess balance was conducted by Clark et al. (2018) In the balance test with Nintendo Wii Balance Board; The participant is asked to complete the 'Basic Balance Test' with their eyes open, within 30 seconds, in 5 stages, with gradually increasing difficulty, using weight transfer to the right and left. The maximum total score that can be obtained from the test is determined as 30.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment Scale. | The assessment will be administered only once to each participant. All tests will be performed on the same day and will take approximately 30 minutes.
  Montreal Cognitive Assessment Scale; In order to distinguish normal individuals from individuals with mild mental problems, Nasreddine et al. (2005). Adaptation of the scale to Turkish was made by Selekler et al. (2010). In this study, the cut-off point of the Turkish version of the scale (21 points) was found to be lower than the original version (26 points).
  The highest score that can be obtained from the scale is 30 and the minimum score is 0.
  In the obtained scores, <10 indicates severe cognitive impairment, 10-17 indicates moderate cognitive impairment, 18-25 indicates mild cognitive impairment, and >26 indicates normal cognition.
  The abbreviation of the scale is "MOCA".
APP- Coo-Test | The assessment will be administered only once to each participant. All tests will be performed on the same day and will take approximately 30 minutes.
  APP-coo-test; It is an application that contains 4 different tests to measure reaction time. The first part consists of 15 white dot tests that test upper extremity coordination, the second part consists of 12 Red Square Tests that test upper extremity speed-coordination, and the third and fourth parts consist of static balance tests. 12 Red Square Tests; It is an application that runs on a touch screen device and can be downloaded from the web for free. It measures the time required to perform the task, in addition, it provides the 12-Red Square Test execution time, average time, standard deviation of trials executed, and coefficient of variation of each upper extremity (dominant and non-dominant hands) at the end of the test. PDF report can be downloaded, printed and signed by the auditor for safekeeping.
Nottingham Health Profile (NIH) | The assessment will be administered only once to each participant. All tests will be performed on the same day and will take approximately 30 minutes.
  Nottingham Health Profile is a quality of life questionnaire, developed in 1975 at the Department of Public Health, University of Nottingham, Faculty of Medicine, England, consisting of two parts, which questions some problems in daily life that require the person to answer himself . The abbreviation of the questionnaire is "NHP".
  Cronbach's α value calculated in all areas of the scale was calculated between 0.56 and 0.83. As a result of the calculations, a result between 0-100 is obtained. A score approaching 100 indicates a low level of perceived health status, and a score approaching 0 indicates a high level of perceived health status.
  The Turkish validity and reliability study of the questionnaire was conducted by Küçükdeveci et al. in 2000.
30 Second Sit and Stand Test | The assessment will be administered only once to each participant. All tests will be performed on the same day and will take approximately 30 minutes.
  30 Second Sit and Stand Test; It is used to evaluate the lower extremity muscle strength and endurance of individuals. At the beginning of the test, individuals are seated on a standard stool with back support, without armrests, approximately 45 cm tall, with their feet flat on the ground and their hands crossed over their shoulders. The test is first demonstrated by a staff member and then administered by a subject. Starting from this position, the patient is asked to sit and stand up as quickly as possible for 30 seconds. The number of times you sit down and stand up correctly for 30 seconds is recorded as the test result. In the literature, the minimum significant difference of the 30-second sit-to-stand test has been determined as 3 repetitions.
Hand Grip Force Test | The assessment will be administered only once to each participant. All tests will be performed on the same day and will take approximately 30 minutes.
  The grip strength test is performed with a dynamometer according to the recommendations of the American Hand Therapists Association. Patients are measured in a sitting position, shoulder adduction, elbow flexion at 90°, forearm prono-supination in neutral and wrist joint in neutral position. 3 consecutive measurements are provided with 60-second rest breaks between measurements. The result obtained from the average of the three measurements is recorded.
Pulmonary Function Test | The assessment will be administered only once to each participant. All tests will be performed on the same day and will take approximately 30 minutes.
  The Pulmonary Function Test is a physiological test that measures airflow or lung volume changes during inspiration and expiration, according to the derivative of time. Its abbreviation is "SFT". Spirometer, on the other hand, is a pulmonary function test device that provides an objective demonstration of the capacity of the lungs and expressed as the percentage of the predicted value according to the guideline of European Respiratory Society (ERS)

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, KAgıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No